CLINICAL TRIAL: NCT05806229
Title: Ultrasound- Guided Mid Point Transverse Process to Pleura Block: Does It Decreases the Incidence of Acute and Chronic Post Nephrectomy Pain? Randomized Controlled Study.
Brief Title: Ultrasound- Guided Mid Point Transverse Process to Pleura Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aliaa Muhammad Belal, LECTURER OF ANESTHESIOLOGY,SURGICAL ICU AND PAIN MEDICINE, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POST NEPHRECTOMY PAIN
Record Dates: First submitted 2023-03-15; First posted 2023-04-10 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Regional Anesthesia for Postnephrectomy Pain
Keywords: nephrectomy pain

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: participants will be masked as they will be under effect of anesthesia while the investigators resposible for pain scoring and clinical assesment are masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): (Mid transverse process to pleura block ) : Patients will receive midpoint transverse process to pleura block with bupivacaine 0.5% (DBK Pharmceutical) (20ml) and dexamethazone 4 mg (SIGMATEC) (1ml) total volume 21 ml
  Interventions: Procedure: Mid transverse process to pleura block (MTP)
- Group II (Sham Comparator): Patients will receive midpoint transverse process to pleura block with 2ml normal saline subcutaneously (shamblock)
  Interventions: Procedure: Mid transverse process to pleura Sham block

INTERVENTIONS:
Procedure: Mid transverse process to pleura block (MTP) — After marking the level of the incision by surgeon (commonly T11 -T12) The patient will be situated in modified lateral position with flank region over kidney elevated to wide the space between iliac crest and subcostal margin, the block area will be sterilized with povidine-iodine, and high -frequency linear ultrasound probe will be placed oblique parasagittally lateral to the spinous process of T11 or T 12 and scanning till appearance of transverse process, 100-mm short bevel echogenic needle (Vygon) will be inserted in plane from cranial to caudal direction. The desired end point of the needle tip will be the midpoint of the line between the posterior border of transverse process and the pleura.After negative aspiration to avoid intravascular injection levobupivacaine 0.5% and dexamethazone 4mg total volume 21ml will be injected
  Arms: Group I
Procedure: Mid transverse process to pleura Sham block — After marking the level of the incision by surgeon (commonly T11 -T12) The patient will be situated in modified lateral position with flank region over kidney elevated to wide the space between iliac crest and subcostal margin, the block area will be sterilized with povidine-iodine, and high -frequency linear ultrasound probe will be placed oblique parasagittally lateral to the spinous process of T11 or T 12 and scanning till appearance of transverse process, 100-mm short bevel echogenic needle (Vygon) will be inserted in plane from cranial to caudal direction. The desired end point of the needle tip will be the midpoint of the line between the posterior border of transverse process and the pleura. with 2ml normal saline subcutaneously will be injected
  Arms: Group II

SUMMARY:
Radical nephrectomy is the surgical process for the resection of malignant tumors of the kidney necessitating a subcostal flank incision.Mild to severe pain is observed in the postoperative period Ineffective pain management leads to several complications. The mid point transverse process to pleura block (MTP) , this technique was used for pain relief after mastectomy, thoracic, abdominal, and spinal surgery and was found effective due to its simplicity and lower risks compared to epidural analgesia.

DETAILED DESCRIPTION:
Ineffective pain management leads to several complications including immobilization, thromboembolism, persisting chronic pain, increased opioid consumption, and delayed hospital discharge.[3]

Multimodal analgesic (MMA) regimens using several drugs and techniques are considered to be necessary for postoperative pain relief. Regional anesthesia techniques, mainly epidural analgesia and more recently, paravertebral blocks became crucial parts of a MMA regimen after the introduction of ultrasound (US) in the regional anesthesia practice.

The mid point transverse process to pleura block (MTP) block was first described as a modified paravertebral block in 2017. The local anesthetic drugs are administered between the transverse process and the pleura. This results in a local anesthetic drugs spread to the dorsal and ventral rami in the paravertebral space through the fenestrations in the superior costotranverse ligament (SCTL) at the level of injection, and frequently to adjacent levels.

This technique was used for pain relief after mastectomy, thoracic, abdominal, and spinal surgery and was found effective due to its simplicity and lower risks compared to epidural analgesia.

ELIGIBILITY:
* Inclusion Criteria: - ASA II and III patients
* scheduled for partial or radical nephrectomy
* standard flank incision either subcostal ,intercostal or supracostal approach
* under general anesthesia.

Exclusion Criteria:

* Bleeding disorders,
* Mental or cognitive dysfunction,
* History of chronic analgesic or drug abuse,
* Allergy to local anesthetics
* Local infection at site of block

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of acute post nephrectomy pain | the first postoperative day
  by Numerical rating score for pain assessment(NRS) minimum value is 0 maximum value is 10 and higher score means poor outcome

SECONDARY OUTCOMES:
chronic post nephrectomy pain development. | the first postoperative 3 monthes
  Numerical rating score for pain assessment (NRS) minimum value is 0 maximum value is 10 and higher score means poor outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Belal, lecturer, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Egypt